CLINICAL TRIAL: NCT00593606
Title: A Phase 3b, Open-Label, Multicenter Trial to Assess the Safety and Tolerability of Switching Korean Subjects From Ropinirole to the Rotigotine Transdermal System and Its Effect on Symptoms in Idiopathic Parkinson's Disease
Brief Title: Safety and Tolerability Trial of Switching From Ropinirole to Rotigotine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0908
Record Dates: First submitted 2007-12-21; First posted 2008-01-15 (Estimated); Results first posted 2009-05-27 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2011-10

CONDITIONS: Parkinson's Disease
Keywords: Rotigotine; NEUPRO; Switching trial from ropinirole to rotigotine,; safety and tolerability; Parkinson disease
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rotigotine (Experimental): Patients were dispensed rotigotine patches up to 8mg/24h at a dose considered by the investigator to be equivalent to the dose of ropinirole that the subject was currently taking.
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Drug: Rotigotine — Strength: 2,4,6,and 8mg/24h, form: transdermal application, once daily application
  Other Names: Neupro

SUMMARY:
This is a Phase 3b, open-label, multicenter trial to assess the safety and tolerability of switching from ropinirole therapy to the rotigotine transdermal system and its effect on symptoms in subjects with idiopathic Parkinson's disease

ELIGIBILITY:
Inclusion Criteria:

* Subject is informed and given ample time and opportunity to think about his/her participation in this trial and has given his/her written informed consent.
* Subject is willing and able to comply with all trial requirements.
* Subject is male or female, aged≥ 18 years.
* Subject is Korean.
* Subjects with idiopathic Parkinson's disease (Hoehn and Yahr Stage I-IV) as defined by the cardinal sign, bradykinesia, and at least 1 of the following: resting tremor, rigidity, or impairment of postural reflexes.
* Subject is not satisfactorily controlled on a total daily dose of ropinirole from 3mg to 12mg, inclusive.
* If the subject is receiving levodopa, either short-acting or sustained-release (in combination with benserazide or carbidopa), the total daily dose must be stable for 28 days prior to the Baseline Visit and must remain stable for the Treatment Period.
* If the subject is receiving an anticholinergic agent (eg, benztropine, trihexyphenidyl, parsitan, procyclidine, biperiden), a monoamine oxidase B (MAO-B) inhibitor (eg, selegiline), a COMT inhibitor (eg, entacapone), or an N-methyl-d-aspartate (NMDA)-antagonist (eg, amantadine), he/she must have been on a stable dose for at least 28 days prior to the Baseline Visit and must be maintained on that dose for the Treatment Period

Exclusion Criteria:

Subjects are not permitted to enroll in the trial if any of the following criteria are met:

* Subject has previously participated in a trial with rotigotine.
* Subject has participated in another trial of an investigational drug within 28 days prior to the Baseline Visit or is currently participating in another trial of an investigational drug.
* Subject has atypical Parkinsonian syndrome(s), including drug-induced Parkinsonian syndrome(s).
* Subject has dementia, active psychosis, or hallucinations (not due to antiparkinsonian medication).
* Subject is receiving therapy with 1 of the following drugs either concurrently or within 28 days prior to Baseline Visit: alpha-methyl dopa, metoclopramide, reserpine, neuroleptics (except specific atypical neuroleptics: olanzapine, ziprasidone, aripiprazole, clozapine, quetiapine), monoamine oxidase A (MAO-A) inhibitors, methylphenidate, or amphetamine.
* Subject is currently receiving central nervous system (CNS) active therapy (eg, sedatives, hypnotics, antidepressants, anxiolytics), unless the dose has been stable for at least 28 days prior to the Baseline Visit and is likely to remain stable for the duration of the trial.
* Subject has a history of seizures or stroke within 1 year, has had a Transient Ischemic Attack (TIA) within 12 months prior to enrollment, or a history of myocardial infarction within the last 6 months prior to enrollment.
* Presence of clinically relevant hepatic dysfunction.
* Presence of clinically relevant renal dysfunction.
* Evidence of clinically relevant cardiovascular disorders.
* Subject has a QTcB interval of ≥ 500ms at Pretreatment or Baseline (repeated measurements within 1 hour).
* Subject has a history of symptomatic (not asymptomatic) orthostatic hypotension in the 6 months prior to Baseline.
* Subject has a history of significant skin hypersensitivity to adhesive or other transdermals or recent unresolved contact dermatitis.
* Subject has malignant neoplastic disease requiring therapy within 12 months prior to enrollment.
* Subject has a history of chronic alcohol or drug abuse within the last 6 months.
* Subject has taken herbal medicine therapy within the last 2 weeks prior to the Baseline Visit.
* Subject has clinically significant laboratory results that, in the judgment of the investigator, would make the subject unsuitable for entry into the trial.
* Subject is pregnant or nursing, or is of childbearing potential but (i) not surgically sterile or (ii) not using adequate birth control methods (including at least 1 barrier method), or (iii) not sexually abstinent or (iv) not at least 2 years postmenopausal.
* Subject has evidence of an impulse control disorder according to the Jay Modified Minnesota Impulsive Disorders Interview (mMIDI) at Pretreatment (Visit 1).
* Subject has any other clinically significant medical or psychiatric condition that would, in the judgment of the investigator, interfere with the subject's ability to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2007-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)

REFERENCES:
- [Result] Kim HJ, Jeon BS, Lee WY, Lee MC, Kim JW, Kim JM, Ahn TB, Cho J, Chung SJ, Grieger F, Whitesides J, Boroojerdi B. Overnight switch from ropinirole to transdermal rotigotine patch in patients with Parkinson disease. BMC Neurol. 2011 Aug 10;11:100. doi: 10.1186/1471-2377-11-100. PMID 21831297
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 124 patients were screened. 5 patients were run-in failures and 3 patients were screen failures. 116 patients started treatment, i.e. were included into the Safety Set. 114 patients were included into the Full Analysis Set. 99 patients completed the treatment period. 2 patients withdrew after the treatment period. 97 patients completed the study.
Period: Overall Study
Arm/Group | Rotigotine
Started | 124
Start of Treatment - Safety Set | 116
Full Analysis Set | 114
Treatment Period Completed | 99
Completed | 97
Not Completed | 27
Not completed — Adverse Event | 13
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 3
Not completed — Lost to Follow-up | 2
Not completed — Run-In Failure | 5
Not completed — Screen Failure | 3

BASELINE CHARACTERISTICS:
Arm/Group | Rotigotine
Number analyzed (Participants) | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 73
  >=65 years | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 47
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 116

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulse Rate (Supine, After 1 Minute)
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
beats per minute | 2.0 (9.4)

2. Primary Outcome: Change in Systolic Blood Pressure (Supine, After 1 Minute)
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
mmHg | 5.7 (14.1)

3. Primary Outcome: Change in Diastolic Blood Pressure (Supine, After 1 Minute)
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
mmHg | 1.7 (9.6)

4. Primary Outcome: Change in Pulse Rate (Supine, After 5 Minutes)
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
beats per minute | 1.8 (8.8)

5. Primary Outcome: Change in Systolic Blood Pressure (Supine, After 5 Minutes)
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 Days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
mmHg | 2.6 (13.1)

6. Primary Outcome: Change in Diastolic Blood Pressure (Supine, After 5 Minutes)
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
mmHg | 0.6 (9.8)

7. Primary Outcome: Change in Pulse Rate (Standing, After 1 Minute)
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
beats per minute | 1.7 (11.8)

8. Primary Outcome: Change in Systolic Blood Pressure (Standing, After 1 Minute)
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
mmHg | -0.2 (12.7)

9. Primary Outcome: Change in Diastolic Blood Pressure (Standing, After 1 Minute)
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
mmHg | 0.8 (10.1)

10. Primary Outcome: Change in Pulse Rate (Standing, After 3 Minutes)
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
beats per minute | 0.8 (11.1)

11. Primary Outcome: Change in Systolic Blood Pressure (Standing, After 3 Minutes)
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
mmHg | 2.0 (12.4)

12. Primary Outcome: Change in Diastolic Blood Pressure (Standing, After 3 Minutes)
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
mmHg | 0.8 (9.1)

13. Primary Outcome: Change in Heart Rate
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
beats per minute | 0.5 (8.7)

14. Primary Outcome: Change in PR Interval
Description: The PR interval is defined as the period that extends from the onset of atrial depolarization (beginning of the P wave) until the onset of ventricular depolarization (beginning of the QRS complex).
  Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Rotigotine
Number analyzed (Participants) | 110
msec | -0.0 (14.6)

15. Primary Outcome: Change in QRS Duration
Description: The QRS duration represents the time it takes for ventricular depolarization to occur.
  Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
msec | -1.2 (6.3)

16. Primary Outcome: Change in QT Interval
Description: The QT interval is the period that extends from the beginning of ventricular depolarization until the end of ventricular repolarization.
  Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
msec | -1.7 (30.5)

17. Primary Outcome: Change in QT Interval Corrected for Heart Rate According to Bazett's Formula (QTcB)
Description: as for outcome 16
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
msec | 0.5 (23.1)

18. Primary Outcome: Change in Percentage of Basophilic Granulocytes in White Blood Cell Count
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: Percentage of white blood cell count
Arm/Group | Rotigotine
Number analyzed (Participants) | 108
Percentage of white blood cell count | 0.01 (0.33)

19. Primary Outcome: Change in Percentage of Eosinophilic Granulocytes in White Blood Cell Count
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: Percentage of white blood cell count
Arm/Group | Rotigotine
Number analyzed (Participants) | 108
Percentage of white blood cell count | -0.11 (1.71)

20. Primary Outcome: Change in Hematocrit
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: l/l*100
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
l/l*100 | 0.09 (1.71)

21. Primary Outcome: Change in Hemoglobin
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: g/l
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
g/l | 0.8 (5.6)

22. Primary Outcome: Change in Percentage of Lymphocytes in White Blood Cell Count
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: Percentage of white blood cell count
Arm/Group | Rotigotine
Number analyzed (Participants) | 108
Percentage of white blood cell count | 0.73 (7.12)

23. Primary Outcome: Change in Percentage of Monocytes in White Blood Cell Count
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: Percentage of white blood cell count
Arm/Group | Rotigotine
Number analyzed (Participants) | 108
Percentage of white blood cell count | 0.96 (8.41)

24. Primary Outcome: Change in Percentage of Neutrophilic Granulocytes Segmented in White Blood Cell Count
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: Percentage of white blood cell count
Arm/Group | Rotigotine
Number analyzed (Participants) | 108
Percentage of white blood cell count | -0.40 (12.69)

25. Primary Outcome: Change in Platelet Count
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: Giga/l
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
Giga/l | 2.6 (29.5)

26. Primary Outcome: Change in Red Blood Cell Count
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: Tera/l
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
Tera/l | 0.023 (0.213)

27. Primary Outcome: Change in White Blood Cell Count
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: Giga/l
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
Giga/l | -0.045 (3.538)

28. Primary Outcome: Change in Albumin
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: g/l
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
g/l | -0.5 (2.1)

29. Primary Outcome: Change in Alkaline Phosphatase
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: Units/l
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
Units/l | -1.4 (16.9)

30. Primary Outcome: Change in Blood Urea Nitrogen
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Rotigotine
Number analyzed (Participants) | 108
mmol/l | -0.24 (1.75)

31. Primary Outcome: Change in Calcium
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
mg/dl | -0.05 (0.30)

32. Primary Outcome: Change in Chloride
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Rotigotine
Number analyzed (Participants) | 108
mmol/l | -0.4 (2.5)

33. Primary Outcome: Change in Creatinine
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
mg/dl | -0.004 (0.101)

34. Primary Outcome: Change in Gamma-Glutamyltransferase
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: Units/l
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
Units/l | -0.1 (7.5)

35. Primary Outcome: Change in Glucose
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
mg/dl | -0.2 (30.0)

36. Primary Outcome: Change in Inorganic Phosphate
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
mg/dl | -0.03 (0.52)

37. Primary Outcome: Change in Potassium
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Rotigotine
Number analyzed (Participants) | 108
mmol/l | 0.08 (0.35)

38. Primary Outcome: Change in Serum Glutamic Oxaloacetic Transaminase
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: Units/l
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
Units/l | -0.1 (7.9)

39. Primary Outcome: Change in Glutamic Pyruvic Transaminase
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: Units/l
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
Units/l | -0.2 (15.6)

40. Primary Outcome: Change in Sodium
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Rotigotine
Number analyzed (Participants) | 108
mmol/l | -0.6 (2.2)

41. Primary Outcome: Change in Total Bilirubin
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
mg/dl | 0.079 (1.133)

42. Primary Outcome: Change in Total Protein
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
g/dl | -0.09 (0.36)

43. Primary Outcome: Change in Uric Acid
Description: Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: µmol/l
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
µmol/l | -3.80 (35.62)

44. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Physical Examination for 'Ears, Eyes, Nose, Mouth, Throat'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 0

45. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Physical Examination for 'Psychiatric'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 0

46. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Physical Examination for 'Hematological/Lymphatic Nodes'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 0

47. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Physical Examination for 'Dermatological'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 1

48. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Physical Examination for 'Cardiovascular'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 0

49. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Physical Examination for 'Peripheral Vascular'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 0

50. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Physical Examination for 'Pulmonary'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 0

51. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Physical Examination for 'Musculoskeletal'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 1

52. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Physical Examination for 'Hepato-/Gastrointestinal'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 0

53. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Physical Examination for 'Renal/Genitourological'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 0

54. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Physical Examination for 'Metabolic/Endocrine'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 0

55. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Physical Examination for 'Other'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 0

56. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Neurological Examination for 'Mental Status'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 0

57. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Neurological Examination for 'Deep Tendon Reflexes'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 0

58. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Neurological Examination for 'Muscle Strength'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 0

59. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Neurological Examination for 'Cranial Nerve Function'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 0

60. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Neurological Examination for 'Plantar Reflex'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 0

61. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Neurological Examination for 'Gait'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 1

62. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Neurological Examination for 'Coordination/Balance'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 0

63. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Neurological Examination for 'Involuntary Movements'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 1

64. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Neurological Examination for 'Sensory Perception'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 0

65. Primary Outcome: Occurrence of Abnormal, Clinically Relevant Events in Neurological Examination for 'Other'
Time Frame: 28 days
Population: Safety Set, only patients with non-missing values were analyzed
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
participants | 0

66. Primary Outcome: Completion of Trial From Baseline to End of Treatment
Time Frame: Baseline, 28 days
Population: Safety Set
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 116
participants | 99

67. Primary Outcome: Completion of Trial on the Original Treatment Assignment From Baseline to End of Treatment
Time Frame: Baseline, 28 days
Population: Safety Set
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 116
participants | 88

68. Primary Outcome: Drop-out During the 5 Half-life Overlap Period Due to Adverse Events (AEs)
Time Frame: Baseline, 2 days
Population: Safety Set
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 116
participants | 0

69. Primary Outcome: Drop-out Due to Adverse Events (AEs) With Onset During the 5 Half-life Overlap Period
Time Frame: Baseline, 56 days
Population: Safety Set
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 116
participants | 9

70. Primary Outcome: Dose Reduction During the 5 Half-life Overlap Period Due to Adverse Events (AEs)
Time Frame: Baseline, 2 days
Population: Safety Set
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 116
participants | 1

71. Primary Outcome: Dose Reduction Due to Adverse Events (AEs) With Onset During the 5 Half-life Overlap Period
Time Frame: Baseline, 56 days
Population: Safety Set
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 116
participants | 1

72. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) Part I Score From Baseline to End of Treatment
Description: The UPDRS is a scale for the assessment of function in Parkinson's disease UPDRS Part I measures 'Mentation, Behavior and Mood'. Range: 0 (Best score possible) to 16 (Worst score possible) Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Full Analysis Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
score on scale | -0.5 (1.2)

73. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) Part II Score From Baseline to End of Treatment
Description: The UPDRS is a scale for the assessment of function in Parkinson's disease UPDRS Part II measures 'Activities in Daily Living'. Range: 0 (Best score possible) to 52 (Worst score possible) Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Full Analysis Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
score on scale | -0.9 (3.3)

74. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) Part III Score From Baseline to End of Treatment
Description: The UPDRS is a scale for the assessment of function in Parkinson's disease UPDRS Part III measures 'Motor Examination'. Range: 0 (Best score possible) to 56 (Worst score possible) Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Full Analysis Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
score on scale | -1.9 (5.9)

75. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) Part IV Score From Baseline to End of Treatment
Description: The UPDRS is a scale for the assessment of function in Parkinson's disease UPDRS Part IV measures 'Complications of Therapy'. Range: 0 (Best score possible) to 23 (Worst score possible) Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Full Analysis Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
score on scale | -0.4 (1.8)

76. Secondary Outcome: Change in Parkinson's Disease Sleep Scale (PDSS) Sum Score From Baseline to End of Treatment
Description: The PDSS is a scale to assess sleep and nocturnal disability in Parkinson's disease.
  Range: 0 (Best score possible) to 60 (Worst score possible) Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Full Analysis Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
score on scale | -0.8 (7.3)

77. Secondary Outcome: Change in Epworth Sleepiness Scale (ESS) Sum Score From Baseline to End of Treatment
Description: The ESS is a self-administered questionnaire in which the subject rates the probability of his/her dozing during 8 situations that are differently conductive to sleep Range: 0 (Best score possible) to 24 (Worst score possible) Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Full Analysis Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 55
score on scale | -0.2 (3.2)

78. Secondary Outcome: Change in Parkinson's Disease Non-Motor Symptom Assessment Scale (PDNMS) Total Sum Score From Baseline to End of Treatment
Description: The PDNMS is a rating by the clinician to assess the severity and frequency of non-motor symptoms in Parkinson's disease patients Range: 0 (Best score possible) to 384 (Worst score possible) Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Full Analysis Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 111
score on scale | -7.9 (19.8)

79. Secondary Outcome: Change in Clinical Global Impression (CGI) Item 1 Score From Baseline to End of Treatment
Description: The CGI is a set of ratings made by a clinician in order to assess the overall severity of an individual's symptoms as well as changes in his/her functioning over time.
  Item 1 measures 'Severity of Parkinson's Disease'. Range: 1 (Normal, not ill at all) to 7 (Among the most extremely ill patients) Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 114
score on scale | -0.0 (0.6)

80. Secondary Outcome: Clinical Global Impression (CGI) Item 2 Score
Description: The CGI is a set of ratings made by a clinician in order to assess the overall severity of an individual's symptoms as well as changes in his/her functioning over time.
  Item 2 measures 'Global Improvement'. Range 1 (Very much improved) to 7 (Very much worse)
Time Frame: 28 days
Population: Full Analysis Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 113
score on scale | 3.6 (1.0)

81. Secondary Outcome: Clinical Global Impression (CGI) Item 3.1
Description: The CGI is a set of ratings made by a clinician in order to assess the overall severity of an individual's symptoms as well as changes in his/her functioning over time.
  Item 3.1 measures 'Therapeutic Effect'. Range: 1 (Marked - Vast improvement. Complete or nearly complete remission of all symptoms.) to 4 (Unchanged or worse)
Time Frame: 28 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 114
participants
  Marked | 3
  Moderate | 20
  Minimal | 36
  Unchanged or Worse | 54
  Not Assessed | 1

82. Secondary Outcome: Clinical Global Impression (CGI) Item 3.2
Description: The CGI is a set of ratings made by a clinician in order to assess the overall severity of an individual's symptoms as well as changes in his/her functioning over time.
  Item 3.2 measures 'Therapeutic Side Effects'. Range: 1 (None) to 4 (Outweigh the therapeutic effect)
Time Frame: 28 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 114
participants
  None | 88
  No Significant Interference with Subj. Functioning | 18
  Significant Interference with Subj. Functioning | 5
  Outweigh the Theraputic Effect | 2
  Not Assessed | 1

83. Secondary Outcome: Patient Global Impression (PGI) Item 1 Score
Description: The PGI is a set of ratings made by the patient in order to assess the overall severity of an individual's symptoms as well as changes in his/her functioning over time.
  Item 1 measures 'Global Improvement'. Range: 1 (Very much improved) to 7 (Very much worse)
Time Frame: 28 days
Population: Full Analysis Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
score on scale | 3.6 (1.2)

84. Secondary Outcome: Patient Global Impression (PGI) Item 2
Description: The PGI is a set of ratings made by the patient in order to assess the overall severity of an individual's symptoms as well as changes in his/her functioning over time.
  Item 2 measures 'Therapeutic Effect'. Range: 1 (Marked - Vast improvement. Complete or nearly complete remission of all symptoms) to 4 (Unchanged or worse)
Time Frame: 28 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 114
participants
  Marked | 5
  Moderate | 25
  Minimal | 38
  Unchanged or Worse | 44
  Missing / Not Done | 2

85. Secondary Outcome: Patient Global Impression (PGI) Item 3
Description: The PGI is a set of ratings made by the patient in order to assess the overall severity of an individual's symptoms as well as changes in his/her functioning over time.
  Item 3 measures 'Side Effects'. Range: 1 (I have no side effects) to 4 (They outweigh the therapeutic effect of the trial medication)
Time Frame: 28 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 114
participants
  No Side Effects | 77
  No Significant Interference with Functioning | 24
  Significant Interference with Functioning | 6
  Outweighing Therapeutic Effect of Trial Medication | 5
  Missing / Not Done | 2

86. Secondary Outcome: Change in Short-form Parkinson's Disease Questionnaire (PDQ-8) Single Index Score From Baseline to End of Treatment
Description: The PDQ-8 is a self-administered 8-item questionnaire that assesses issues associated with Parkinson's disease.
  Range: 0 (good health) to 100 (poor health) Change = 28 day value minus baseline value.
Time Frame: Baseline, 28 days
Population: Full Analysis Set, only patients with non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 112
score on scale | -3.9 (13.5)

87. Secondary Outcome: Patient Treatment Preference Scale Question 1
Description: Have you used pharmaceutical treatments for your Parkinson's disease before the study?
Time Frame: 28 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 114
participants
  yes | 114
  no | 0

88. Secondary Outcome: Patient Treatment Preference Scale Question 2
Description: Why did you decide to enter this study?
Time Frame: 28 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 114
participants
  Side effects with oral medicine | 14
  Oral medicine not effective in controlling sympt. | 21
  Taking med. several times a day was not convenient | 71
  Other | 40

89. Secondary Outcome: Patient Treatment Preference Scale Question 3
Description: In comparing the patch and previous oral treatments for Parkinson's disease, how satisfied have you been with oral medication / patch?
Time Frame: 28 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 114
participants
  Very Dissatisfied with Oral Medication | 3
  Dissatisfied with Oral Medication | 11
  Neither Satisfied nor Dissatisfied with Oral Med. | 49
  Satisfied with Oral Medication | 43
  Very Satisfied with Oral Medication | 6
  Assessment for Oral Medication Missing / Not Done | 2
  Very Dissatisfied with Patch | 9
  Dissatisfied with Patch | 28
  Neither Satisfied nor Dissatisfied with Patch | 34
  Satisfied with Patch | 32
  Very Satisfied with Patch | 9
  Assessment for Patch Missing / Not Done | 2

90. Secondary Outcome: Patient Treatment Preference Scale Question 4
Description: I would prefer using a patch over taking a pill or capsule for treatment of my Parkinson's disease.
Time Frame: 28 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 114
participants
  Strongly Agree | 18
  Agree | 34
  Neither Agree nor Disagree | 29
  Disagree | 28
  Strongly Disagree | 3
  Not Done / Missing | 2

91. Secondary Outcome: Patient Treatment Preference Scale Question 5
Description: I would prefer applying one 40cm**2 patch over applying two 20cm**2 patches for treatment of my Parkinson's disease.
Time Frame: 28 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 114
participants
  Strongly Agree | 17
  Agree | 68
  Neither Agree nor Disagree | 10
  Disagree | 13
  Strongly Disagree | 4
  Not Done / Missing | 2

92. Secondary Outcome: Patient Treatment Preference Scale Question 6
Description: What aspects do you like the most about the patch?
Time Frame: 28 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 114
participants
  Applying the patch once a day | 81
  Comfortable to wear | 28
  Does not interfere with my normal activities | 61
  Do not have to take medicine in public | 56
  Provides symptom relief all day | 46
  Convenient | 53
  Easy to apply | 50
  Do not have to remember to take med. during day | 60
  Missing / Not Done | 2

93. Secondary Outcome: Patient Treatment Preference Scale Question 7
Description: What aspects do you like the least about the patch? Check all that apply.
Time Frame: 28 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 114
participants
  Hard to apply | 11
  Hard to remove | 3
  Hard to remove the patch from its pouch | 1
  Did not stay on for the entire day | 80
  Uncomfortable to wear | 27
  Not always covered by clothing | 8
  Symptom relief did not last all day | 29
  Not Done / Missing | 2

ADVERSE EVENTS:
Arm/Group | Rotigotine
Serious Adverse Events (participants affected / at risk) | 0/116
Other Adverse Events (participants affected / at risk) | 45/116
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=116)
Dry Mouth (Gastrointestinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 6 (7)
Fatigue (General disorders) | 2 (2)
Application site pruritus (General disorders) | 3 (3)
Pain (General disorders) | 2 (2)
Gait disturbence (General disorders) | 1 (2)
Oedema peripheral (General disorders) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyskinesia (Nervous system disorders) | 6 (6)
Bradykinesia (Nervous system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 7 (7)
Dizziness postural (Nervous system disorders) | 1 (2)
Tremor (Nervous system disorders) | 7 (8)
Somnolence (Nervous system disorders) | 4 (4)
Parkinson's disease (Nervous system disorders) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Rapid eye movements sleep abnormal (Psychiatric disorders) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1)
Libido increased (Psychiatric disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.